CLINICAL TRIAL: NCT06431152
Title: Administration of sEV Derived From UC-MSC in Patients With Osteoarthritis of the Knee: Safety Determination in a Pilot Dose-escalation Study
Brief Title: Intra-articular Injection of UC-MSC Exosome in Knee Osteoarthritis
Acronym: EXO-OA01
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Universidad de los Andes, Chile (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EXO-OA01
Record Dates: First submitted 2024-05-17; First posted 2024-05-28 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Osteo Arthritis Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Low-Dose (Experimental): Intra-articular knee injection of exosomes (2 x 10e9 particles/dose) derived from allogeneic mesenchymal stromal cells. Single dose.
  4 patients
  Interventions: Biological: UC-MSC sEV
- Medial-Dose (Experimental): Intra-articular knee injection of exosomes (6 x 10e9 particles/dose) derived from allogeneic mesenchymal stromal cells. Single dose.
  4 patients
  Interventions: Biological: UC-MSC sEV
- High-Dose (Experimental): Intra-articular knee injection of exosomes (2 x 10e10 particles/dose) derived from allogeneic mesenchymal stromal cells. Single dose.
  4 patients
  Interventions: Biological: UC-MSC sEV

INTERVENTIONS:
Biological: UC-MSC sEV — Small extracellular vesicles derived from allogenic mesenchymal stromal cells, single dose
  Other Names: Cellistem®sEV-OA

SUMMARY:
The study aim to evaluate safety of exosomes (sEVs) from allogeneic mesenchymal stromal cells delivered by an intra-articular injection in the knee of patients with mild to moderate symptomatic osteoarthritis. The sEVs will be produced in a GMP-facility. The investigators expect to enroll 12 patients in this phase 1 trial open label dose-escalation pilot and the follow-up will be up to 12 months.

DETAILED DESCRIPTION:
The clinical investigation will represent a Phase 1 trial focusing on small extracellular vesicles derived from mesenchymal stem cell (MSC-sEV) in patients with symptomatic Kellgren II-III knee OA. The phase 1 component of the study will be an open-label dose escalation pilot study in which three cohorts of subjects with OA will receive increasing doses of UC-MSC-sEV administered as a single intra-articular (IA) injection. Each cohort will comprise four participants. Eligible study subjects will be enrolled at the "Clinica Universidad de los Andes".

The small extracellular vesicles derived from umbilical cord mesenchymal stem cell (UC-MSC-sEV) will be prepared in the "Clinica Universidad de los Andes" GMP facility. The sEV-based therapeutic for clinical use will be manufactured in compliance with standardized procedures based on Good Manufacture Practice (GMP) regulations and all quality controls aforementioned. The sEV therapeutic will be transported to the patient administration site under controlled conditions, ensuring maintenance of a temperature range between 2-8°C. The sEV injection is expected to be administered within the first 6 h of product manufacture.

The primary study endpoints of this trial will focus on the safety, feasibility, and toxicity of the sEV-based product. The phase I will examine (1) the incidence of immediate post-infiltration adverse reactions in patients; (2) the occurrence of synovitis post-infiltration in patients at 24 and 48 hours, as well as on days 7 and 15; (3) the frequency of post-infiltration pain reported by patients at 24 and 48 h, and on days 7 and 15; and (4) the prevalence of adverse events related to sEV therapy occurring beyond IA infiltration at 24 and 48 h, and on days 7 and 15, as well as at months 2, 4, 6, 8, 10, and 12. The secondary study endpoint will be determine the optimal dose for phase II trials. The criteria that will be considered are (1) Safety profile at infiltration at 24 and 48 h, and on days 7 and 15, as well as at months 2, 4, 6, 8, 10, and 12; (2) changes in WOMAC scores at months 2, 4, 6, 8, 10, and 12; and (3) alterations in the Visual Analog Scale (VAS) pain scores at months 2, 4, 6, 8, 10, and 12.

ELIGIBILITY:
Inclusion Criteria:

* Age 30 to 70 years.
* Kellgren-Lawrence grade II - III knee OA (Rosenberg view x-ray)
* VAS for pain ≥ 40 mm, without surgical indication in the affected knee.
* In case of bilateral involvement, the most affected knee will be treated. The contralateral knee should be asymptomatic or present a VAS ≤ 20 mm.
* Stable knee with normal physical examination.
* Signed Informed Consent

Exclusion Criteria:

* Symptomatic bilateral knee OA
* BMI > 30 kg/m2
* Joint instability at physical examination.
* Mechanical meniscal tear on physical examination.
* Associated conditions: active local or systemic infection, neoplasia, immunosuppression, pregnancy, anticoagulant therapy, coagulation disorders, inflammatory joint disease (autoimmune, by crystal or other), joint prosthesis, symptomatic spine or hip disease.
* Recent use of intra-articular (last 6 months) or oral (last month) steroid therapy.
* Recent use of intra-articular hyaluronic acid therapy (last 6 months)
* Subchondral bone fracture.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Adverse Event | 12 month
  Occurrence of any adverse reactions within 12 months of treatment

SECONDARY OUTCOMES:
Incidence of injection-related pain according to Visual Analogue Scale (VAS) (0-100mm) | 1-2 weeks
  Pain measured by Visual Analogue Scale (VAS) (0-100mm) after first week of treatment
Incidence of injection-related synovitis according to effusion grading scale of knee joint | 1-2 weeks
  Synovitis measured by effusion grading scale (zero to 3+) after first week of treatment
Pain change | 12 months
  Change in Visual Analogue Scale (VAS) (0-100mm) score every 2 months
Disability change | 12 months
  Change in WOMAC subscale (Western Ontario and McMaster Universities Osteoarthritis IndexWomac) related to function (C) every 2 months Pain (0-20), Stiffness (0-8), functional capacity (0-68).
Percentage of responders | 52 weeks
  According to OMERACT-OARSI Criteria Index Response after 52 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Clinica Universidad de los Andes, Santiago, Las Condes, Chile

IPD SHARING:
Plan to Share IPD: No